CLINICAL TRIAL: NCT03340974
Title: An Adaptive Phase I/II Dose Escalation Trial of Stereotactic Body Radiation Therapy in Combination With Radiomodulating Agent GC4419 in Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Pilot Dose Escalation Trial of Stereotactic Body Radiation Therapy (SBRT) in Combination With GC4419 in Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI-4419-101
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Stereotactic Body Radiation Therapy
Keywords: Avasopasem manganese
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — avasopasem manganese; Radiosurgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GC4419 90mg +50 Gy SBRT (Experimental): Avasopasem manganese (GC4419) +SBRT
  Interventions: Drug: GC4419; Radiation: Stereotactic Radiation Therapy (SBRT) 50 Gy
- GC4419 90 mg + 55 Gy SBRT (Experimental): Avasopasem manganese (GC4419) +SBRT
  Interventions: Drug: GC4419; Radiation: Stereotactic Radiation Therapy (SBRT) 55 Gy
- Placebo + 50 Gy SBRT (Placebo Comparator): Placebo +SBRT
  Interventions: Drug: Placebo; Radiation: Stereotactic Radiation Therapy (SBRT) 50 Gy
- Placebo + 55 Gy SBRT (Placebo Comparator): Placebo + SBRT
  Interventions: Drug: Placebo; Radiation: Stereotactic Radiation Therapy (SBRT) 55 Gy

INTERVENTIONS:
Drug: GC4419 — 90 mg Avasopasem (GC4419) per day daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT to assigned dose level
  Other Names: Avasopasem manganese
  Arms: GC4419 90 mg + 55 Gy SBRT; GC4419 90mg +50 Gy SBRT
Drug: Placebo — Placebo daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT to assigned dose level
  Arms: Placebo + 50 Gy SBRT; Placebo + 55 Gy SBRT
Radiation: Stereotactic Radiation Therapy (SBRT) 50 Gy — Dose-finding will be done using the sequentially adaptive phase I-II Late onset Efficacy-Toxicity (LO-ET) trade-off-based design.
  Arms: GC4419 90mg +50 Gy SBRT; Placebo + 50 Gy SBRT
Radiation: Stereotactic Radiation Therapy (SBRT) 55 Gy — Dose-finding will be done using the sequentially adaptive phase I-II Late onset Efficacy-Toxicity (LO-ET) trade-off-based design.
  Arms: GC4419 90 mg + 55 Gy SBRT; Placebo + 55 Gy SBRT

SUMMARY:
The purpose of the phase I/II clinical study is to determine the best dose of fractionated stereotactic radiation therapy (SBRT) given either with Avasopasem manganese (GC4419) or placebo to patients who have been diagnosed with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a parallel arm adaptive design phase I-II dose-finding study to determine the optimal dose of fractionated stereotactic radiation therapy (SBRT), given either with the radiomodulating agent Avasopasem manganese (GC4419) or placebo for treatment of locally advanced pancreatic cancer. Dose-finding will be done using the sequentially adaptive phase I-II Late onset Efficacy-Toxicity (LO-ET) trade-off-based design [1-3].

A maximum of 48 patients will be randomized 1:1 to Arm A or Arm B. Patients in Arm A will receive Avasopasem manganese (GC4419) in combination with their assigned SBRT dose, and patients in Arm B will receive Placebo (PBO) with their assigned SBRT dose. The randomization will be restricted so that the sample size within each arm is exactly 24 patients.

GC4419/placebo will be given intravenously in a one hour infusion. SBRT must be initiated as soon as possible upon completion of the GC4419/placebo infusion.

GC4419/placebo will be given beginning on the first day of radiation and continuing daily, concurrent M-F throughout the administration of SBRT

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or biopsy confirmed adenocarcinoma of the pancreatic head, body or tail
2. Disease that is appropriate for SBRT by virtue of being:

   a. Locally advanced and technicallyunresectable, as determined by a pancreaticobiliary surgeon as part of a multidisciplinary review at the investigative site, including multi-phasic CT demonstrating: i.Greater than 180 degree tumor involvement of the superior mesenteric artery ii. Greater than 180 degree tumor involvement of the celiac axis, including major branches of the celiac axis that render it unresectable (e.g. common hepatic artery).

   iii. Tumor involvement of the first branch of the SMA that is not surgically reconstructible iv. Long segment involvement of the superior mesenteric vein/portal vein or hepatic artery that is not surgically reconstructible b. Potentially resectable, but patient is judged not a candidate for surgery, after multidisciplinary review at the investigative site; c. Potentially resectable, but the patients refuses surgery and is considered an acceptable candidate for SBRT after multidisciplinary review at the investigative site; d. "Borderline" resectable, as determined by multidisciplinary review, including absence of distant lymphadenopathy and the primary tumor characterized by one of more of the following: i. A tumor-vessel interface (TVI) with the mesenteric vein (SMV) or portal vein (PV) measuring ≥180° of the circumference of either vein's wall or short-segment occlusion of either vein with a normal vein above or below the obstruction amenable to reconstruction; ii. Any TVI with the common hepatic artery (CHA) with normal artery proximal and distal to the TVI amenable to reconstruction; iii. A TVI with the superior mesenteric artery (SMA) measuring <180° of the circumference of the vessel wall
3. Pancreatic tumor size and limited bowel involvement by tumor must be judged acceptable for SBRT at the discretion of the treating investigator
4. No evidence of distant metastasis either prior to or after induction chemotherapy.
5. Completion of at least 3 months of standard induction chemotherapy for LAPC, which should consist of either FOLFIRINOX, gemcitabine or nab-paclitaxel or another standard combination of induction chemotherapy agents
6. Patient must have metal stent in place if duodenal stent is required. If patient has plastic stent, this must be replaced prior to radiation.
7. Ability to understand and follow the breathing instructions involved in the respiratory gating procedure or to tolerate compression sufficient to reduce fiducial motion to <= 5mm.
8. Age 18 years or older
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (0, 1 or 2)
10. Adequate hematologic function as indicated by i. Absolute neutrophil counts (ANC) ≥ 1,500/mm3 ii. Hemoglobin (Hgb) ≥ 8.0 g/dL iii. Platelet count ≥ 75,000/mm3
11. Adequate renal and liver function as indicated by:

    i. Creatinine ≤ 1.5 x upper-normal limit (ULN) ii. Total bilirubin ≤ 1.5 x upper-normal limit (ULN) iii. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN iv. Alkaline phosphatase ≤ 2.5 x ULN
12. Properly obtained written informed consent

Exclusion Criteria:

1. Prior radiation therapy to the abdomen that would overlap with treatment field
2. Prior surgical resection of pancreatic tumor
3. Receiving any approved or investigational anti-cancer agent other than those provided for in this study
4. Uncontrolled or active gastric or duodenal ulcer disease within 30 days of enrollment
5. Visible invasion of tumor into the lumen of the bowel or stomach on endoscopy (Note: Radiological infiltration into bowel is allowed, unless deemed clinically unsafe.)
6. Residual or ongoing ≥ Grade 3 non-hematologic toxicity from chemotherapy
7. Contraindication to IV contrast
8. Concurrent participation in another interventional clinical trial or use of another investigational agent within 30 days of study entry Note: Patients who are participating in non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would limit compliance with treatment
10. Second primary malignancy within the last 5 years, unless treated definitively and with low risk of recurrence in the judgment of the treating investigator
11. Known history of HIV or active hepatitis B/C (patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible)
12. Female patients who are pregnant or breastfeeding
13. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for 30 days after the last dose of GC4419. This includes any woman who has experienced menarche but has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH levels greater than 35 mIU/mL. A negative urine or serum pregnancy test must be obtained within 14 days prior to the start of study therapy in all women of child-bearing potential.
14. Male subjects who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 90 days after the last dose of GC4419 are excluded.
15. Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure.
16. Medical history that includes any condition, or requires the use of concomitant medications which, in the investigator's judgment, are associated with or create a risk of increased carotid sinus sensitivity, symptomatic bradycardia, or syncopal episodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kennedy, MD, Study Chair — Galera Therapeutics
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoffe S, Frakes JM, Aguilera TA, Czito B, Palta M, Brookes M, Schweizer C, Colbert L, Moningi S, Bhutani MS, Pant S, Tzeng CW, Tidwell RS, Thall P, Yuan Y, Moser EC, Holmlund J, Herman J, Taniguchi CM. Randomized, Double-Blinded, Placebo-controlled Multicenter Adaptive Phase 1-2 Trial of GC 4419, a Dismutase Mimetic, in Combination with High Dose Stereotactic Body Radiation Therapy (SBRT) in Locally Advanced Pancreatic Cancer (PC). Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1399-1400. doi: 10.1016/j.ijrobp.2020.09.022. Epub 2020 Nov 18. No abstract available. PMID 33427657
- [Derived] Taniguchi CM, Frakes JM, Aguilera TA, Palta M, Czito B, Bhutani MS, Colbert LE, Abi Jaoude J, Bernard V, Pant S, Tzeng CD, Kim DW, Malafa M, Costello J, Mathew G, Rebueno N, Koay EJ, Das P, Ludmir EB, Katz MHG, Wolff RA, Beddar S, Sawakuchi GO, Moningi S, Slack Tidwell RS, Yuan Y, Thall PF, Beardsley RA, Holmlund J, Herman JM, Hoffe SE. Stereotactic body radiotherapy with or without selective dismutase mimetic in pancreatic adenocarcinoma: an adaptive, randomised, double-blind, placebo-controlled, phase 1b/2 trial. Lancet Oncol. 2023 Dec;24(12):1387-1398. doi: 10.1016/S1470-2045(23)00478-3. PMID 38039992
- [Derived] Sishc BJ, Ding L, Nam TK, Heer CD, Rodman SN, Schoenfeld JD, Fath MA, Saha D, Pulliam CF, Langen B, Beardsley RA, Riley DP, Keene JL, Spitz DR, Story MD. Avasopasem manganese synergizes with hypofractionated radiation to ablate tumors through the generation of hydrogen peroxide. Sci Transl Med. 2021 May 12;13(593):eabb3768. doi: 10.1126/scitranslmed.abb3768. PMID 33980575

RESULTS

PARTICIPANT FLOW:
Groups:
- GC4419 90 mg +50 Gy SBRT: 90 mg Avasopasem manganese (GC4419) per day daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT (50 Gy)
- GC4419 90 mg +55 Gy SBRT: 90 mg Avasopasem manganese (GC4419) per day daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT (55 Gy)
- Placebo + 50 Gy SBRT: Placebo daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT (50 Gy)
- Placebo +55 Gy SBRT: Placebo daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT (55 Gy)
Period: Active Protocol Treatment
Arm/Group | GC4419 90 mg +50 Gy SBRT | GC4419 90 mg +55 Gy SBRT | Placebo + 50 Gy SBRT | Placebo +55 Gy SBRT
Started | 18 | 6 | 6 | 12
Completed (Completed 12 month Follow up Period) | 18 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Completion of Study -Long Term Follow up
Arm/Group | GC4419 90 mg +50 Gy SBRT | GC4419 90 mg +55 Gy SBRT | Placebo + 50 Gy SBRT | Placebo +55 Gy SBRT
Started | 18 | 6 | 6 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 18 | 6 | 6 | 12
Not completed — Death | 8 | 5 | 5 | 7
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — Last Know Alive | 8 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- GC4419 90 mg +50 Gy; GC4419 90mg +55 Gy: Avasopasem (GC4419) + SBRT
  GC4419: 90 mg Avasopasem (GC4419) per day daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT to assigned dose level
- Placebo +50 Gy; Placebo +55 Gy: Placebo +SBRT
  Placebo: Placebo daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT to assigned dose level
- Total: Total of all reporting groups
Arm/Group | GC4419 90 mg +50 Gy | GC4419 90mg +55 Gy | Placebo +50 Gy | Placebo +55 Gy | Total
Number analyzed (Participants) | 18 | 6 | 6 | 12 | 42
Age, Customized [Count of Participants; unit: Participants]
  Age group (years): Age Group 18-65 years | 4 | 2 | 3 | 4 | 13
  Age group (years): Age Group 66-75 | 8 | 3 | 1 | 8 | 20
  Age group (years): Age Group >75 | 6 | 1 | 2 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 6 | 19
  Male | 13 | 3 | 1 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 2 | 5
  Not Hispanic or Latino | 14 | 6 | 6 | 9 | 35
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 3
  White | 16 | 5 | 4 | 12 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 6 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: CTCAE Grade 3 or 4 Gastro-intestinal (GI) Toxicities or Death Within 90 Days From the Start of Therapy
Description: Number of Common Terminology Criteria Adverse Events (CTCAE) that are grade 3 or 4 gastro-intestinal (GI) toxicities or deaths. CTCAE grade 3 or 4 gastro-intestinal toxicities are those adverse events that a subject may experience in their gastro-intestinal system that have been graded by the treating investigator to be severe (Grade 3) or life-threatening (Grade 4).
Time Frame: Within 90 days from the start of therapy "related" after CTCAE
Population: Intent-to-Treat (ITT) population, which consisted of all randomized subjects who received at least 1 dose of GC4419/placebo and/or SBRT. The ITT population excluded randomization failures (ie, randomized subjects who did not receive any GC4419/placebo or SBRT).
Measure: Number; unit: Events
Groups:
- GC4419 90 mg + 50 Gy: SBRT + Avasopasem (GC4419)
  GC4419: 90 mg Avasopasem (GC4419) per day daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT .
- GC4419 90 mg +55 Gy: SBRT + Placebo
  Placebo: Placebo daily (60 min IV infusion, prior to SBRT), concurrent with daily fractions of SBRT to assigned dose level
Arm/Group | GC4419 90 mg + 50 Gy | GC4419 90 mg +55 Gy | Placebo + 50 Gy SBRT | Placebo +55 Gy SBRT
Number analyzed (Participants) | 18 | 6 | 6 | 12
Events
  Deaths within 90 days from last dose of study treatment | 1 | 0 | 0 | 0
  Grade 3 or 4 Gastrointestinal Toxicities | 1 | 1 | 0 | 1

2. Primary Outcome: Radiographic Stable Disease (SD) or Better Based on RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST) criteria for target lesions that are assessed by radiographic imaging : Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the longest diameter of the target lesions; Stable disease (SD) is neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for local progressive disease (LPD); Local Progressive Disease (LPD) is at least a 20% increase in the longest diameter of the target lesion, utilizing the baseline measurement as reference.
Time Frame: All subjects assessed with at least 12 months of follow up following the administration of SBRT
Population: Intent-to-Treat (ITT) population which consisted of all randomized subjects who received at least 1 dose of avasopasem/placebo and/or SBRT with the most restrictive censoring scenario ( subjects censored at the time of surgery, new anti-cancer therapy, and new malignancy)
Measure: Count of Participants; unit: Participants
Arm/Group | GC4419 90 mg +50 Gy | GC4419 90mg +55 Gy | Placebo +50 Gy | Placebo +55 Gy
Number analyzed (Participants) | 18 | 6 | 6 | 12
Participants
  Stable Disease | 12 | 3 | 5 | 8
  Partial Response | 4 | 3 | 1 | 1
  Progressive Disease | 0 | 0 | 0 | 1
  Not Evaluated/Censored | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of subject randomization until 12 months following the last dose of SBRT (total duration approximately 14 months)
Arm/Group | GC4419 90 mg +50 Gy | GC4419 90mg +55 Gy | Placebo +50 Gy | Placebo +55 Gy
All-Cause Mortality (participants affected / at risk) | 8/18 | 5/6 | 5/6 | 7/12
Serious Adverse Events (participants affected / at risk) | 7/18 | 1/6 | 0/6 | 4/12
Other Adverse Events (participants affected / at risk) | 9/18 | 5/6 | 6/6 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 90 mg +50 Gy (N=18) | GC4419 90mg +55 Gy (N=6) | Placebo +50 Gy (N=6) | Placebo +55 Gy (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 90 mg +50 Gy (N=18) | GC4419 90mg +55 Gy (N=6) | Placebo +50 Gy (N=6) | Placebo +55 Gy (N=12)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (5) | 4 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 1 (1) | 3 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (3) | 1 (1) | 2 (2)
Blood alkaline phosphatase increase (Investigations) | 2 (5) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 3 (4) | 3 (5) | 5 (7) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Erucation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3) | 4 (4)
Pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 2 (4) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the proposed study manuscript for publication, presentation or other disclosure must first be forwarded to Sponsor not less than 30 days prior to submission for review and comment. PI agrees to delete or revise references to confidential information upon Sponsor's request and PI agrees to to consider all other comments of Sponsor in good faith.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03340974/Prot_SAP_000.pdf